CLINICAL TRIAL: NCT07053254
Title: The Characteristics and Treatment Mechanism of Vascular Grafts in Elderly Patients With CAOD Through Single-cell Transcriptome Analysis
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-0197
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Occlusive Disease (CAOD)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fixed tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to establish a cardiovascular biobank using vascular grafts obtained from participants with coronary artery occlusive disease (CAOD). Through genomic and transcriptomic analyses, the study seeks to characterize the biological features of the vascular grafts and identify potential therapeutic targets and mechanisms related to vascular remodeling and stiffness.

DETAILED DESCRIPTION:
This observational study will utilize discarded vascular graft tissues obtained during coronary artery bypass grafting (CABG) procedures in participants with coronary artery occlusive disease (CAOD). Our surgical team performs over 200 CABG operations annually, allowing for the consistent and ethical acquisition of excess graft tissue without requiring any additional procedures or interventions for participants.

Collected tissues will be processed as follows:

A portion of each graft will be preserved in RNAlater solution for molecular analyses, including total RNA sequencing, quantitative PCR, and western blotting.

Another portion will be fixed in formalin and embedded for histological examination, including immunohistochemistry (IHC), to validate mechanisms of vascular remodeling and stiffness at the protein level.

This approach ensures that all biological samples are collected with minimal risk and no additional burden to participants, while enabling comprehensive multi-omic analysis to investigate the pathophysiological characteristics of vascular grafts in elderly CAOD patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older, Patients scheduled to undergo coronary artery bypass grafting (CABG), Patients who voluntarily provide written informed consent for study participation, Patients who are able and willing to comply with study procedures during the study period

Exclusion Criteria:

* Pediatric or adolescent patients under 18 years of age, Patients requiring concomitant surgical correction for valvular heart disease, Patients undergoing reoperative (redo) cardiac surgery, Patients who decline to provide informed consent prior to surgery

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender Eligibility Description: All sexes are eligible to participate. Both male and female patients undergoing coronary artery bypass grafting (CABG) will be included.
Study Population: Participants will include adult patients diagnosed with coronary artery occlusive disease (CAOD) who are undergoing elective or urgent coronary artery bypass grafting (CABG). Vascular graft tissues (e.g., internal mammary artery or saphenous vein) that are not required for anastomosis and would otherwise be discarded during surgery will be collected for molecular and histological analysis. No additional procedures or interventions will be performed on participants beyond standard clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2027-04-11 (Estimated); Study Completion 2027-04-11 (Estimated)

PRIMARY OUTCOMES:
Identification of gene expression profiles associated with vascular stiffness in graft tissues | At the time of surgery (single timepoint sample collection)
  To identify differentially expressed genes and signaling pathways related to vascular stiffness using total RNA sequencing of vascular graft tissues obtained during coronary artery bypass grafting (CABG).

SECONDARY OUTCOMES:
Validation of stiffness-related gene targets and correlation with clinical and histological parameters | Within 2 year after tissue collection
  To validate selected stiffness-associated gene targets identified through RNA sequencing using qPCR and western blotting; to assess corresponding protein expression through immunohistochemistry; and to correlate transcriptomic findings with participants' clinical characteristics such as age, hypertension, and diabetes.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiovascular Surgery, Severance Cardiovascular Hospital , Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No